CLINICAL TRIAL: NCT04947787
Title: Establishing a Physical Activity Referral Scheme for People With Noncommunicable Diseases in the German Healthcare System
Acronym: BewegtVersorgt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Klaus Pfeifer, Head of the Department of Sport Science and Sport, University of Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BewegtVersorgt
Record Dates: First submitted 2021-06-09; First posted 2021-07-01 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Non-Communicable Chronic Diseases
Keywords: physical activity promotion; physical activity referral scheme; physician-initiated; behaviour change
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants receive a physical activity referral scheme.
  Interventions: Behavioral: Physical activity referral scheme (PARS)
- Control Group (Active Comparator): Participants receive physical activity advice from general practitioners.
  Interventions: Behavioral: Physical activity advice (PAA)

INTERVENTIONS:
Behavioral: Physical activity referral scheme (PARS) — Participants of the intervention group will receive brief physician advice and be referred to an exercise professional (e.g., physiotherapist, sports therapist) for a more intensive counseling intervention. The counseling intervention consists of an initial assessment, individual physical activity counseling (360'), a final assessment after 12 weeks, and a follow-up assessment after 24 weeks.
  Arms: Intervention Group
Behavioral: Physical activity advice (PAA) — Participants of the control group will only receive brief physician advice regarding the promotion of physical activity and as an information sheet with tips on how to adopt a more physically active lifestyle.
  Arms: Control Group

SUMMARY:
The BewegtVersorgt project involved co-producing a physical activity referral scheme (PARS) for inactive persons with underlying non-communicable diseases. Various relevant actors of the German healthcare system (e.g., representatives of physicians, health insurance providers, sports organizations, exercise representatives of exercise professions, representatives of patients) participated in the co-production process.

The purpose of this study is to evaluate the effectiveness of co-produced PARS in the Erlangen-Nuremberg-Fürth region. Local general practitioners and exercise professionals will carry out the implementation of the PARS in standard care. The cluster-randomized study includes two intervention arms; one group will receive specific support from physical activity experts to increase physical activity (PARS). The control group will receive only the physician's advice and then continue to engage in physical activity on their own (PAA). The participants will be followed up at 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older; living in the region of Erlangen-Nürnberg-Fürth, Germany;
* At least one of the following existing non-communicable diseases (controlled type 2 diabetes mellitus; cardiovascular diseases; obesity (BMI ≥ 30 kg/m2); arthrosis in knee and/or hip);
* Not meeting German PA recommendations (less than 150 minutes/week of moderate-intensity aerobic activity or less than 75 minutes/week of vigorous-intensity aerobic activity or any other equivalent combination);
* The person can safely participate in physical activities based on general practitioners' clinical judgment.

Exclusion Criteria:

* The person plans to leave the region of Erlangen-Nürnberg-Fürth during the study period;
* The person participating in another study with similar content;
* The person is or plans to be absent for more than four weeks during the 12-week-intervention period;
* Person has cognitive impairments that prevent an effective communication with the general practitioner and the therapist;
* Persons with mental illness such as psychotic, substance abuse, mood, personality disorders;
* Unstable clinical situation or serious health impairments that prevent from undertaking physical activity safely (e.g., acute myocardial infarction, unstable angina pectoris, fever, terminal tumor diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in self-reported moderate to vigorous physical activity (min/week): BSA 3.0 questionnaire | Baseline (T0), 12 weeks (T1), and 24 weeks (T2)
  The Physical Activity, Exercise, and Sport Questionnaire (Bewegungs- und Sportaktivität Fragebogen; BSA-F) is a German questionnaire that assesses the amount of physical activity during the last four weeks. It differentiates between leisure-time/transportation activities (physical activity score) and sport-/exercise-related activities (sports score). Participants are required to report the frequency and duration of activities executed during the last four weeks. Minutes of leisure-time physical activity per week and sport-/exercise-related activity per week are calculated to get the physical activity and the sports score. Both scores can be combined to receive the overall volume of physical activity completed during leisure-time/transportation and sport-/exercise-related activities.
Changes in physical activity-related health competence: BGK Questionnaire | Baseline (T0), 12 weeks (T1), and 24 weeks (T2)
  This will be measured by the German version of the Physical Activity-Related Health Competence questionnaire. The questionnaire consists of 44 total items that measure three sub-competencies necessary for a health-promoting physical activity behavior: movement competence (20 items; min = 0, max = 17.6), control competence (10 items; min = 0, max = 10.8), physical activity-related self-regulation competence (14 items; min = 0, max = 14.8). Higher scores indicate higher competencies.

SECONDARY OUTCOMES:
Changes in quality of life: EuroQol (EQ-5D-5L) | Baseline (T0), 12 weeks (T1), and 24 weeks (T2)
  The EQ-5D-5L is a self-administered quality of life scale that consists of a descriptive system and a visual analog scale. The descriptive system contains five well-being dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Each dimension has five levels of severity (no problems, slight problems, moderate problems, severe problems, unable to/extreme problems), each coded with numbers from one to five. The result obtained is a 5-digit code that represents the health state profile of the participant. The visual analog scale assesses the overall current health.
Changes in self-efficacy towards physical activity: Selbstwirksamkeit zur sportlichen Aktivität-Skala (SSA-Scale) | Baseline (T0), 12 weeks (T1), and 24 weeks (T2)
  This will be measured by a German instrument (Selbstwirksamkeit zur sportlichen Aktivität; SSA-Scale), including 12 items that assess the confidence someone has to perform a planned physical activity in the face of various conditions that may act as barriers. Each item is scored on a seven-point Likert scale representing the level of confidence from '1' meaning not sure at all and '7' meaning the participant is very confident of performing the physical activity as planned even in the face of a particular challenge. The total scores range from 12 to 84, where the higher the score, the greater the self-efficacy.
Changes in participants' perceived autonomy support: Health Care Climate Questionnaire-Deutschland (HCCQ-D) | Baseline (T0), 24 weeks (T1; only intervention group)
  We will use the German version of the Health Care Climate Questionnaire (HCCQ-D) to measure the participant's perception of autonomy support from the general practitioner. It incorporates 15 statements with seven-point response options that indicate the level of agreement ranging from strongly disagree to strongly agree. Higher scores indicate higher perceived autonomy support.
Changes in stages of change: transtheoretical model (TTM) | Baseline (T0), 12 weeks (T1), and 24 weeks (T2)
  We will use one German question that is based on the transtheoretical model of behavior change. The five response options represent five stages of change: pre-contemplation, contemplation, preparation, action, and maintenance.
Changes in sport- and movement-related self-concordance: Sport- und bewegungsbezogenen Selbstkonkordanz Skala (SSK-Scale) | Baseline (T0), 12 weeks (T1), and 24 weeks (T2)
  This will be evaluated with the self-administered German scale (Sport- und bewegungsbezogenen Selbstkonkordanz-Skala; SSK-Scale) that measures the self-concordance. The SSK-Scale contains 12 items grouped into four subscales: intrinsic, identified, introjected, and extrinsic motivation. The subscales' scores for introjected and extrinsic motivation will be subtracted from the sum of the identified and intrinsic motivation subscales to receive the overall score. Thus, the overall score ranges from minus ten (-10) to ten, where a higher score suggests a higher level of sports- and movement-related self-concordance.

OTHER OUTCOMES:
Experience of participating actors (general practitioners, exercise professionals): (semi-) structured interviews | Through study completion, an average of 1 year
  The (semi-) structured interview is based on RE-AIM and asks specifically about adoption, implementation, and maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Pfeifer, Prof. Dr., Principal Investigator — Friedrich-Alexander-University Erlangen-Nürnberg
Locations (1):
- Friedrich-Alexander-University Erlangen-Nürnberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Klamroth S, Mino E, Naber I, Weissenfels A, Geidl W, Gelius P, Abu-Omar K, Pfeifer K. Coproducing a physical activity referral scheme in Germany: a qualitative analysis of stakeholder experiences. BMJ Open. 2024 May 22;14(5):e082710. doi: 10.1136/bmjopen-2023-082710. PMID 38777585
- [Derived] Weissenfels A, Klamroth S, Carl J, Naber I, Mino E, Geidl W, Gelius P, Abu-Omar K, Pfeifer K. Effectiveness and implementation success of a co-produced physical activity referral scheme in Germany: study protocol of a pragmatic cluster randomised trial. BMC Public Health. 2022 Aug 13;22(1):1545. doi: 10.1186/s12889-022-13833-2. PMID 35964042